CLINICAL TRIAL: NCT01838460
Title: Elevated Dose of Sublingual Nicotine Tablets Compared With Swedish Snus. Nicotine Pharmacokinetics and Subjective Effects of Single Doses.
Brief Title: Sublingual Nicotine Tablets Compared With Swedish Snus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Contract Research Organization el AB (Industry)
Collaborators: Commitum AB (Industry)
Responsible Party: Principal Investigator, Erik Lunell, MD, PhD, Medical Director, Contract Research Organization el AB
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SM WS 12
Record Dates: First submitted 2013-02-19; First posted 2013-04-24 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Tobacco, Smokeless

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- 6 mg dose of sublingual nicotine tablets (Experimental): 6 mg dose of sublingual nicotine tablets, single dose.
  Interventions: Drug: sublingual nicotine tablets
- PSWM 0.5 g (16 mg nicotine/g) (Active Comparator): Swedish portion snus, smokeless tobacco, PSWM 0.5 g (16 mg nicotine/g), single dose
  Interventions: Other: Smokeless tobacco
- PSWL 1.0 g (8 mg nicotine /g) (Active Comparator): Swedish portion snus, smokeless tobacco, PSWL 1.0 g (8 mg nicotine /g), single dose
  Interventions: Other: Smokeless tobacco
- PSWL 1.0 g (16 mg nicotine /g) (Active Comparator): Swedish portion snus, smokeless tobacco, PSWL 1.0 g (16 mg nicotine /g), single dose
  Interventions: Other: Smokeless tobacco
- PSWL (8 mg nicotine /g) 2x1.0 g (Active Comparator): Swedish portion snus, smokeless tobacco, PSWL (8 mg nicotine /g) 2x1.0 g, single dose
  Interventions: Other: Smokeless tobacco

INTERVENTIONS:
Drug: sublingual nicotine tablets — 6 mg = 3 tablets
  Other Names: Nicorette Sublingual Tablets
  Arms: 6 mg dose of sublingual nicotine tablets
Other: Smokeless tobacco — Swedish type moist snuff
  Other Names: PSWM 0.5 g; PSWL 1.0 g
  Arms: PSWL (8 mg nicotine /g) 2x1.0 g; PSWL 1.0 g (16 mg nicotine /g); PSWL 1.0 g (8 mg nicotine /g); PSWM 0.5 g (16 mg nicotine/g)

SUMMARY:
To compare each subject's AUCinf, after administration of one single dose of 6 mg of Nicorette sublingual nicotine tablets ( three 2mg tablets) to that of one single 1 g dose of SS containing 16 mg nicotine.

DETAILED DESCRIPTION:
Open, randomized, five-way cross-over. Single dose administration. The Nicorette 6 mg sublingual tablets and three strengths of SS are tested. Subjects are 18-50 years old, male/female (non-pregnant), healthy volunteer, using minimum 12 pouches of 1 g portion snus or half a can of loose snus per day. The treatments are given as single doses in randomized order. The subject keeps the sublingual tablets still under the tongue for 30 minutes.

The subject keeps the pouch(es) of snus still between the upper lip and the gum for 30 minutes. Serial blood samples are drawn before, and at regular time intervals up to 6 hours after administration.

Amount of nicotine extracted, plasma nicotine concentration at 30 minutes (C30), Tmax, Cmax, AUCinf and heart rate for each treatment. The AUCinf area is based on plasma data corrected for background nicotine (time zero sample).

Each subject's rating of subjective effects using a Visual Analogue Scale (VAS) on a palm top computer, anchored with "not at all" to "extremely".

VAS scores will be obtained at the plasma concentrations sampling time points up to 30 minutes for:

* craving intensity
* overall "product strength" (head rush, "buzz", "hit", feeling alert)
* increased salivation
* burning sensation in the mouth and/or throat

ELIGIBILITY:
Inclusion Criteria:

1. Consent to participate voluntarily and sign Informed Consent Form prior to any study procedure.
2. Healthy male/female, age 18 through 50 years. Female using contraceptive pill or negative pregnancy test.
3. Willing and able to comply with study procedures.
4. Snus user, minimum 12 pouches or half a can of loose snus per day of pouched portion snus, minimum 1 gram/portion.
5. Abstinent from any form of nicotine use from 8.00 p.m.
6. Fasting overnight from 11.00 p.m.

Exclusion Criteria:

1. Smoker, defined as "smoking during the last 24 hours according to self report and CO in exhaled air >10 ppm at clinical visits"
2. Second or third degree AV block or sick sinus syndrome; congestive heart failure classified as functional Class III or IV by the New York Heart Association; myocardial infarction within six months of baseline; a prolonged QTc interval at screen or pretreatment (defined as a QTc interval of > 450 msec for males or > 470 msec for females); other clinically significant heart conditions which would negatively impact on the subject completing the study.
3. Subjects with clinically significant liver disease which may prevent the subject from completing the study and/or an elevation in total bilirubin, alkaline phosphatase, LDH, ASAT, or ALAT of > 3 times the upper limit of the laboratory reference interval.
4. Subjects with clinically significant renal disease which may prevent the subject from completing the study and/or an elevation in serum creatinine of > 1.5 times the laboratory reference.
5. Surgery within 6 months of the Baseline visit that, in the opinion of the investigator, could negatively impact on the subject's participation in the clinical study.
6. Subjects who have participated in other drug studies within 30 days prior to enrolment.
7. Subjects with any surgical or medical condition, which, in the judgment of the clinical investigator, might interfere with the absorption, distribution, metabolism or excretion of the drug.
8. Subjects who are using drugs capable of inducing hepatic enzyme metabolism within the previous 30 days (or 5 half lives of inducing agent, whichever is longer) of enrolment in this study.
9. Subjects with a medical history of seizures.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
AUCinf | 6 hours

SECONDARY OUTCOMES:
craving intensity | 6 hours
head rush | 6 hours
  overall "product strength" (head rush, "buzz", "hit", feeling alert
burning sensation | 6 hours
  burning sensation in the mouth and/or throat
increased salivation | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Erik Lunell, Md, Phd, Principal Investigator — Croel AB
Locations (1):
- Carema Specialistvård, Eslöv, Eslöv, Skåne County, Sweden